CLINICAL TRIAL: NCT07008690
Title: Magnetic Resonance Imaging of the Temporomandibular Joint in Patients With Degenerative Joint Disease
Brief Title: MRI of the TMJ in Patients With DJD
Status: Active, not recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: University of Minnesota - DJD
Record Dates: First submitted 2025-05-28; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Degenerative Joint Disease; Control Subjects
Keywords: Degenerative joint disease; TMJ; MRI; Controls; Healthy controls; Magnetic resounance imaging; Diagnosis
MeSH Terms: conditions — Joint Diseases; Disease | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (2):
- DJD: Participants must be 18 years or older, who can attend a 2-hour MRI appointment at the CMRR. They must have a clinically confirmed diagnosis of degenerative joint disease (DJD) based on CT, radiographs, or traditional MRI.
  Interventions: Diagnostic Test: MRI
- Controls: Participants must be 18 years or older who can attend a 2-hour MRI appointment at the CMRR. They must confirm the absence of any pre-existing temporomandibular joint (TMJ) disease.
  Interventions: Diagnostic Test: Magnetic Resonance Imaging

INTERVENTIONS:
Diagnostic Test: MRI — This exploratory study will longitudinally image patients diagnosed with DJD, capturing multiple bilateral TMJ MRI scan images over the course of 18 months using 3T MRI.
  Groups: DJD
Diagnostic Test: Magnetic Resonance Imaging — For comparison, this exploratory study will image patients that are not diagnosed with DJD, capturing multiple bilateral TMJ MRI scan images over the course of 4 weeks.
  Groups: Controls

SUMMARY:
This observational research is comparative in design, that is assessing the change in qMRI measures in degenerative changes of the TMJ in patients diagnosed with DJD. These patients will be imaged multiple times over the course of 18 months, using clinical 3T MRI scanners located at the Center for Magnetic Resonance Research (CMRR), and their findings will be compared to controls; individuals who are not diagnosed with DJD. No investigational agents or MRI contrast agents will be used.

DETAILED DESCRIPTION:
Participants with DJD will be recruited during routine examinations at the TMD clinic located at the School of Dentistry, UMN. They will be approached by their clinicians for potential enrollment in an MRI study. Eligibility will be assessed based on prior imaging and medical history. If eligible and interested, participants will complete a consent process and a CMRR questionnaire which is a safety screening questionnaire, followed by scheduling for a 2-hour MRI session at the CMRR. During the visit, participants will undergo approximately 90 minutes of qMRI scans using a 15-channel face coil. Afterward, they'll complete an exit questionnaire. Additional follow-up scans may occur over 18 months, following the same procedures, while control participants will have two scans 1-4 weeks apart.

ELIGIBILITY:
Inclusion Criteria:

1. To participate in this study, patients (with DJD) must:

   * Be 18 years or older
   * Provide written informed consent in English
   * State willingness to comply with all study procedures and be available for the duration of the study
   * Have clinically confirmed DJD diagnoses based on CT and/or radiographs, and /or traditional MRI scan obtained by their clinician.
   * Willing to have a separate approximately 2-hour appointment to have an MRI at the CMRR
   * Has the ability to manage their own calendar and schedule appointments
   * Does not have a serious medical condition
   * Is not pregnant or is not potentially pregnant
2. To participate in this study, controls (participants without DJD) must:

   * Be 18 years or older
   * Provide written informed consent in English
   * State willingness to comply with all study procedures and be available for the duration of the study
   * Confirm the absence of any pre-existing TMJ disease
   * Willing to have a separate approximately 2-hour appointment to have an MRI at the CMRR
   * Has the ability to manage their own calendar and schedule appointments
   * Does not have a serious medical condition
   * Is not pregnant or is not potentially pregnant
3. Exclusion Criteria:

Participants will be excluded if they:

* Contraindications to MRI. Exclusion criteria for MRI are:

  1. Ferromagnetic implants
  2. History of shrapnel or shot gun injury
  3. Too large to fit in the magnet (body mass index >= 40, approx.)
  4. Cardiac pacemakers
  5. Severe claustrophobia
  6. Large tattoos
  7. History of metalwork
* Are non-English speaking
* Could be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with DJD will be recruited during routine examinations at the TMD clinic located at the School of Dentistry, UMN. If eligible and interested, participants will undergo approximately 90 minutes of qMRI scans. Additional follow-up scans may occur over 18 months, while control participants will have two scans 1-4 weeks apart.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-11-28 (Estimated)

PRIMARY OUTCOMES:
Assess the change in qMRI measures in degenerative changes of the TMJ over time | 1.5 year
  We will assess these changes between baseline MRI and multiple MRI scanning session over the course of 18 months. We will group patients who do (case group) and do not (control group) have clinical progression of DJD based on their existing CT scans and/or radiograph imaging acquired by their clinician to confirm their diagnosis. These findings will be evaluated through subjective observations and the ability to identify various anatomical structures. Additionally, intra- and inter-rater reliability analyses will be conducted to assess the consistency of the MRI interpretations

SECONDARY OUTCOMES:
Build a rich MRI data set | 1.5 years
  This exploratory study is designed to provide useful data regardless of the outcomes. This study will begin to build a rich MRI data set that will lay the groundwork for future, larger studies to more fully evaluate the quantitative MRI techniques and address important clinical questions.

CONTACTS AND LOCATIONS:
Locations (1):
- Orofacial MRI Center at UMN, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No